CLINICAL TRIAL: NCT05193084
Title: MONITORED-HF: Remote MONIToring Of Ambulatory intRavEnous Diuretics in Heart Failure
Brief Title: Remote Monitoring of Ambulatory Intravenous Diuretics in Heart Failure
Acronym: MONITORED-HF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heartfelt Technologies (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: MRI01
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Oedema; Heartfelt Device
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Work Stream 1 (WS1): The general aim of this work stream is to assess the hypothesis "can the volumes measured by the Heartfelt device be useful in titrating and optimising drug management for patients undergoing home-IV diuretics and after completion of IV-diuretic treatment.?"
  We will characterise the data collected by the Heartfelt device in the participants' home, correlating it to weight readings (either from the scales or paper weight diary) and medical observations recorded while patients are being treated with IV Diuretics.
  Patients from WS1 will be invited to keep the device in their home for 3 months in total, which will therefore cover periods during which they do not receive IV diuretics, but are still at relatively high risk of decompensation. That data will be analysed in the same fashion as the data collected in WS2.
  Interventions: Device: Heartfelt Device; Device: Connected weighing scales
- Work Stream 2 (WS2): The general aim of WS2 is to assess the hypothesis "can the Heartfelt device be used to monitor heart failure stability and detect fluid overload in patients recently discharged after an episode of decompensated heart failure?".
  This work stream will also aim to examine whether the Heartfelt device gives an indication of the number of days prior to hospital admissions that the Heartfelt device can detect changes in foot volume. This will be achieved by comparing the data collected by the Heartfelt device in the participants' home, and correlating it to weight readings and medical observations. Hospital admissions will be a particularly useful correlation point as it would provide information on the detection of the forming oedema leading up to this event. In future, the information collected during this study will be used to design and power an interventional study to demonstrate the effectiveness of such data in providing a leading indicator of hospitalisation.
  Interventions: Device: Heartfelt Device; Device: Connected weighing scales

INTERVENTIONS:
Device: Heartfelt Device — The Heartfelt Device is a CE marked device that measures the volume of the foot/lower leg. By positioning the Heartfelt device in the bedroom, automatic measurements can be made whenever the subject gets in and out of bed. Feet identification software, complemented by manual checks, ensures that photographs are only taken of the specified subject. Data is censored so that the part of the body which is 50cm above the floor is not stored. Encrypted, anonymised data is transmitted over the internet to the company's secure servers. For this study, no personal identifiable data will be stored on the device or on the servers used by the device.
  The volume readings collected can be presented to the clinical team on a web interface. This is not presented against identifiable data, but only participant ID. However, in the current pilot, volume readings will not be reviewed by the clinical team until the point of data analysis, after the study period.
Device: Connected weighing scales — The connected weighing scales are Xiaomi Smart Scales (CE marked, manufactured by Anhui Huami Informeyshn Technologies).
  The participant will be instructed to use those scales for the period of the study, as often as directed by their healthcare professional(s) (the fact that a participant has not used scales regularly in the past is not an exclusion criteria). The weighing scales display weight so that the participants can record the weight in their own heart failure records (paper weight diary).
  The study team will check the patient's paper weight diary in case they choose to use another set of scales.
  The participant will be able to see the weight readings on the weighing scales during the study.
  The scales will record patient weight as well as the date and time of the measurements.

SUMMARY:
This study will aim to collect proof of concept data to inform the study design of a larger paired comparison study to establish key research questions about the Heartfelt device. The current study will be run with 2 parallel workstreams. Both are presented here:

Data collected from Work Stream 1 (WS1) is expected to give an indication of the usefulness of the volumes measured by the Heartfelt device in optimising diuretic therapy for patients undergoing ambulatory-IV diuretic treatment, as well as looking at the usefulness of foot volume changes monitoring post IV Diuretic treatment. As these patients are often managed in a home / community setting, objective indicators to assess oedema during treatment are currently limited.

Data collected from Work Stream 2 (WS2), patients recently discharged after a heart failure hospitalisation (HFH), is expected to determine if the Heartfelt device can be used to monitor heart failure stability and detect fluid overload in patients recently discharged from hospital after an episode of decompensated heart failure. The investigators may also be able to get an indication of the number of days prior to hospital admission during which the Heartfelt device can detect changes in foot volume.

Both workstreams will provide qualitative feedback, from health care practitioners, patients and carers in both groups about their experience using the Heartfelt Device.

DETAILED DESCRIPTION:
Heart failure hospitalisations are common, but some are potentially preventable through early detection and timely optimisation of pharmacotherapies, most often diuretic titration.

Peripheral oedema is a cardinal feature of heart failure decompensation, though not all patients seek medical attention at this time. The detection of this increase in volume may therefore be a useful tool in preventing heart failure decompensation and hospitalisation.

This study will evaluate a completely automated (no contact) device which captures volumes of the patient's feet in their home, with the ultimate aim of this data being accessible to the heart failure team. However for the purpose of this study, the clinical team will be blinded to the data in order to be able to assess the temporal relationship (and time) between an alert being generated by the device and a hospital admission, or medication change. However if for example a patient fall is detected by the device, a designated Manchester clinician can be contacted to act.

Peripheral oedema is a cardinal feature of heart failure decompensation, though not all patients seek medical attention at this time. The detection of this increase in volume may therefore be a useful tool in preventing heart failure decompensation and hospitalisation.

In WS1 of the current study, the investigators will specifically be looking at whether the use of the Heartfelt Technology can be used to support the remote monitoring of clinical response to home-based intravenous(IV) diuretic interventions as part of an admission avoidance strategy. Our hypothesis is that the Heartfelt technology coupled with this home intervention could provide clinically useful objective measurement of peripheral oedema, which could be used by the heart failure team to titrate the diuretics and guide duration of treatment.

This pilot study will examine change in longitudinal volumes measured by the device and home IV diuretic dosage as well as daily clinical observations. This will help confirm the validity of the readings provided by the device.

Once the home-based intravenous(IV) diuretic intervention is complete, patients will continue to be monitored for a total of 3 months, to observe relative stability or detect further clinically significant decompensations.

In WS2 of the current study, the investigators will be looking at whether Heartfelt alert can offer a window of opportunity in which to perform a theoretical clinical intervention. In order to establish the lead time, recently discharged patients, a population known to be at high risk of re-admission, will be provided with the Heartfelt device and a post-hoc analysis of the data will be performed to establish the number of days between the alert being raised by the Heartfelt device and the date of diagnosis of decompensation +/- hospital admission where this occurs.

This study will be a small-scale pilot to collect information which will support the set-up of a larger study. The pilot will be purely observational as the investigators will not intervene based on the Heartfelt readings. The post-hoc analysis will be undertaken to inform the design of the larger study. As soon as a patient has had the device disconnected, their data can be reviewed for analysis as their participation in the study is completed at that point. This may allow for preliminary analysis to be completed part way through the wider study.

During the pilot the investigators will also collect acceptability ratings from patients and carers.

Research in Heart failure has been reported to often recruit non representative patient groups (Younger patients generally and fewer women and BAME patients than expected for example). So the investigators plan to compare data from the study participants to the ones of the overall HF population seen at the hospital (already recorded as part of the NICOR records). The demographic that the investigators plan to compare are: deprivation level (from postcode), age, sex and ethnicity.

ELIGIBILITY:
Work stream 1 Inclusion Criteria:

1. Patient is willing and able to provide written informed consent.
2. Diagnosis of heart failure
3. Patient with peripheral oedema requiring IV diuretics
4. Patient accepted for co-management by the MFT Heart Failure and home IV team*

   * There may be some instances where the patient is under the management of the MFT HF team but attends the day unit for IVs due to capacity or other logistical considerations. These patients can also be enrolled in the evaluation.

Work stream 1 Exclusion Criteria:

1. Patient has bandages to lower limbs everyday
2. Patient has an amputation of the foot
3. Patient lacks capacity to consent
4. Patient is not ambulant or unable to mobilise unaided around the house
5. Patient is of no fixed abode
6. Patient has potentially reversible cause of decompensated heart failure and is awaiting intervention (revascularisation/ valvular intervention)
7. Patient taking part in a conflicting evaluation/study that could confound the results of this evaluation by and/or impact clinical interventions and patient outcomes
8. Patient must not be pregnant, and is taking relevant birth control if of child-bearing potential*

Note that a patient not able to comply with daily weights is NOT an exclusion criteria as the Heartfelt Device should provide data for these patients despite their lack of ability to adhere to the usual monitoring protocol.

*Note that criteria (h) has been requested by the insurance for clinical trial cover. However we do not expect participants of this study to be trying to get pregnant (the typical age of patients is expected in an earlier evaluation was around 70 years ).

Work stream 2 Inclusion Criteria:

1. Patient is willing and able to provide written informed consent.
2. Diagnosis of heart failure
3. Patient under follow up with the MFT HF service
4. Patient with a recent admission with decompensated heart failure in last 12 months OR who received home IV diuretics within the last 12-months
5. Patient has been discharged on at least furosemide 80mg or equivalent diuretic dose

Work stream 2 Exclusion Criteria:

1. Patient has bandages everyday
2. Patient has an amputation of the foot
3. Patient lacks capacity to consent
4. Patient is not ambulant or unable to mobilise unaided around the house
5. Patient is of no fixed abode
6. Patient has potentially reversible cause of decompensated heart failure and is awaiting intervention (revascularisation/ valvular intervention)
7. Patient taking part in a conflicting evaluation/study that could confound the results of this evaluation by increasing clinic workload burden for that patient and/or impact clinical interventions and patient outcomes
8. Patient must not be pregnant, and is taking relevant birth control if of child-bearing potential*

Note that a patient not able to comply with daily weights is NOT an exclusion criteria as the Heartfelt Device should provide data for these patients despite their inability to use weighing scales at times.

*Note that criteria (h) has been requested by the insurance for clinical trial cover. However we do not expect participants of this study to be trying to get pregnant (the typical age of patients is expected in an earlier evaluation was around 70 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be aged 18 years or older with a diagnosis of heart failure at the time of signing the informed consent form and be under the care of the Heart Failure service at Manchester University NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Use of the device to optimise drug management | 3 months
  Can the volumes measured by the Heartfelt device be useful in titrating and optimising drug management for patients undergoing home-IV diuretics? (WS1)
Use of the device to monitor heart failure stability and detect fluid overload | 3 months
  Can the Heartfelt device can be used to monitor heart failure stability and detect fluid overload in patients recently discharged after an episode of decompensated heart failure? (WS2)
Response to device by patients | 3 months
  Is the device well received by patients?
Response to device by carers | 3 months
  Is the device well received by carers?

SECONDARY OUTCOMES:
Number of days prior to hospital admission the device can detect changes in foot volume | 3 months
  Examine whether the Heartfelt device gives an indication of the number of days prior to hospital admissions that the Heartfelt device can detect changes in foot volume (WS2).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fozia Ahmed, MBChB, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- The Manchester Heart Centre Manchester University NHS Foundation, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided